CLINICAL TRIAL: NCT00766844
Title: Cervical Spinal Cord Stimulation for the Prevention of Cerebral Vasospasm Following Aneurysmal Subarachnoid Hemorrhage Using MTS Trial System 3510
Brief Title: Cervical Spinal Cord Stimulation for the Prevention of Cerebral Vasospasm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Konstantin V. Slavin (Other)
Responsible Party: Sponsor-Investigator, Konstantin V. Slavin, Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UIC 2007-0899; FDA IDE G060177/S001 (Other: FDA)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: vasospasm; spinal cord stimulation; aneurysm; subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active (Experimental): Spinal cord stimulation
  Interventions: Device: spinal cord stimulation

INTERVENTIONS:
Device: spinal cord stimulation — electrode is inserted into cervical epidural space for continuous spinal cord stimulation

SUMMARY:
The study investigates safety, feasibility and effectiveness of cervical spinal cord stimulation (SCS) in prevention of cerebral arterial vasospasm following aneurysmal subarachnoid hemorrhage (aSAH).

It is postulated that 2 week long stimulation of the cervical spinal cord using an implanted epidural electrode will prevent or decrease severity of cerebral arterial vasospasm following aSAH.

DETAILED DESCRIPTION:
Continuous stimulation of the cervical spinal cord for 14 days after electrode implantation (within 3 days after aneurysmal subarachnoid hemorrhage). The single-arm single-institution non-randomized prospective study evaluates effects of cervical spinal cord stimulation on prevention of cerebral arterial vasospasm.

The patients are followed for 12 months after completion of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Subarachnoid hemorrhage (SAH) within 72 hours
* Ruptured aneurysm confirmed by angiography of CT angiography
* Fisher grade 2-4
* Hunt & Hess grade 2-4
* Aneurysm is secured
* Ability to obtain informed consent

Exclusion Criteria:

* Pregnancy
* Allergy to IV contrast or to any component of SCS system
* Non-aneurysmal SAH
* Previous cervical spine surgery or any anomaly of cervical spine that would prevent electrode insertion
* Coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Prevention of cerebral vasospasm | 14-17 days after aSAH

SECONDARY OUTCOMES:
Any complication of spinal cord stimulation | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin V Slavin, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center in Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Slavin KV, Vannemreddy P. Cervical spinal cord stimulation for prevention and treatment of cerebral vasospasm after aneurysmal subarachnoid hemorrhage: clinical and radiographic outcomes of a prospective single-center clinical pilot study. Acta Neurochir (Wien). 2022 Nov;164(11):2927-2937. doi: 10.1007/s00701-022-05325-4. Epub 2022 Aug 3. PMID 35920945